CLINICAL TRIAL: NCT02536521
Title: Study on the Predictive Variables Able to Predict the Hemodynamic Effect of Intra-abdominal Pressure in the Children Undergoing Laparoscopic Surgery
Brief Title: Predictive Variables of the Hemodynamic Effect During the Laparoscopic Surgery in Children
Acronym: Lapa-BP
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Other Study IDs: H-1507-039-686
Record Dates: First submitted 2015-08-24; First posted 2015-09-01 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Laparoscopic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Hemodynamically stable
- Hemodynamically unstable: Hemodynamically unstable patients are defined as those with a 20% decrease in systolic blood pressure according to the change of intraabdominal pressure.

SUMMARY:
This prospective observational study aimed to identify the intraoperative variables to predict the hemodynamic change according to intra-abdominal pressure in the children undergoing laparoscopic surgery.

The intraoperative variables includes Pulse pressure variation (PPV), systolic pressure variation (SPV), stoke volume variation (SVV), Pulse oximeter plethysmographic waveform amplitude (△POP),and pleth variability index (PVI).

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients undergoing laparoscopic surgery

Exclusion Criteria:

* known arrhythmia
* known lung disease
* known cardiac dysfunction (Ejection fraction less than 30%)

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients undergoing laparoscopic surgery
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2015-08; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Pleth variability index(PVI) | Outcome measure will be assessed before the CO2 desufflation for about 2minutes.

SECONDARY OUTCOMES:
Systolic pressure variation(SPV) | Outcome measure will be assessed before the CO2 desufflation for about 2minutes.
Pulse pressure variation(PPV) | Outcome measure will be assessed before the CO2 desufflation for about 2minutes
Pulse oximeter plethysmographic waveform amplitude (△POP) | Outcome measure will be assessed before the CO2 desufflation for about 2minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim EH, Lee JH, Song IK, Ryu HG, Kim HS, Kim JT. Assessment of dynamic variables of fluid responsiveness to predict desufflation-induced hypotension during paediatric laparoscopic surgery. Br J Anaesth. 2017 Nov 1;119(5):956-963. doi: 10.1093/bja/aex172. PMID 28981568